CLINICAL TRIAL: NCT01826539
Title: A Comparison of Dorsal Branch of the Digital Nerve Versus Dorsal Digital Nerve for Finger Pulp Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TSChen8652; HBTS13-03095 (Other: Ethics Committee of Hebei)
Record Dates: First submitted 2013-04-01; First posted 2013-04-08 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Soft Tissue Defect of the Finger
Keywords: Dorsal digital nerve; dorsal branch of the digital nerve; dorsal branch of the digital artery; dorsal digital island flap; finger pulp defect.

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Innervated finger flap (Other): donor nerve attached with the flap for finger pulp reconstruction
  Interventions: Procedure: flap includes a donor nerve

INTERVENTIONS:
Procedure: flap includes a donor nerve — the donor nerve is attached with the flap for sensory reconstruction of the finger

SUMMARY:
As the donor nerve attached with the flap, the dorsal branch of the digital nerve and the dorsal digital nerve is commonly used for finger pulp reconstruction.This study compares two donor nerves: the dorsal branch of the digital nerve and the dorsal digital nerve.

DETAILED DESCRIPTION:
The investigators compares two donor nerves attached with the flap for sensory reconstruction of finger pulp: the dorsal branch of the digital nerve and the dorsal digital nerve. The main outcomes were static 2-point discrimination and Semmes-Weinstein monofilament scores of the flap, and pain and cold intorlence of the reconstructed finger.

ELIGIBILITY:
Inclusion Criteria:

* The pulp or fingertip defect in only one finger
* A defect greater than or equal to 1.5 cm in length
* Necessity to preserve finger length
* A patient between 18 and 60 years of age

Exclusion Criteria:

* Injuries to the dorsum of the middle phalanx
* Injuries to the course of the vascular pedicle or donor nerve
* A defect less than 1.5 cm in length
* Multiple finger pulp defect
* Extremely contaminated wounds

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
static 2-point discrimination (2PD) test | 18 months to 26 months
  The test points are at the center of the radial or ulnar portion of the pulp. Each area is tested 3 times with a Discriminator. We stop at 4mm as a limit of 2PD and consider this normal.

SECONDARY OUTCOMES:
Cold intolerance | 18 months to 26 months
  Cold intolerance in the reconstructed finger is assessed using the self-administered Cold Intolerance Severity Score questionnaire [10]. The maximum score is 100 and was group into 4 ranges (0-25, 26-50, 51-75, and 76-100), corresponding to mild, moderate, severe, and extreme severity, respectively.

OTHER OUTCOMES:
Pain | 18 months to 26 months
  Using the visual analogue scale (VAS), patients are asked to report pain sensations of the reconstructed pulps and donor sites. The VAS consists of a 10 cm line that is grouped into mild (0-3 cm), moderate (4-6 cm) and severe (7-10 cm).

CONTACTS AND LOCATIONS:
Overall Officials: Dequn Liu, MD. PhD, Study Director — The Second Hospital of Tangshan
Locations (1):
- The Second Hospital of Tangshan, Tangshan, Hebei, China

REFERENCES:
- [Result] Chen C, Tang P, Zhang X. Use of the dorsal digital sensate free flap for reconstruction of volar soft tissue defect of digits. Ann Plast Surg. 2014 May;72(5):537-41. doi: 10.1097/SAP.0b013e318268a97f. PMID 23241796